CLINICAL TRIAL: NCT06274866
Title: Investigation Of The Effects Of A Home Based Exercise Program Under Physiotherapist Supervision Following Total Hip Arthroplasty And Comparison With The Control Group
Brief Title: Effects Of A Home Based Exercise Program Following Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: dsahinoglu
Record Dates: First submitted 2024-02-02; First posted 2024-02-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: PHYSİOTHERAPY
Keywords: Total Hip Arthroplasty; Home Based Exercise Program; Balance; Pain; Function
MeSH Terms: conditions — Pain | interventions — Resistance Training; Control Groups

STUDY DESIGN:
Intervention Model Description: Randomize controlled two groups
Masking Description: no blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): After total hip arthroplasty, participants who take supervised home based exercised program which consists especially early weight bearing hip specific mobilization and strengthening exercises.
  Interventions: Other: exercise program
- Control group (Other): After total hip arthroplasty, participants who take an educational booklet (about exercise program) at hospital stay
  Interventions: Other: control group

INTERVENTIONS:
Other: exercise program — Study group were followed up with a personalized home-based exercise program for 6 weeks. IThe exercise program of the individuals in the study group was checked at two-week intervals and adjustments were made in the exercise program
  Other Names: educational supervised exercises
  Arms: Study Group
Other: control group — Individuals in the control group were followed up with an exercise training brochure.
  Other Names: educational booklet
  Arms: Control group

SUMMARY:
The aim of this study is to examine the effects of home-based exercise on pain-related factors, postural control and early functional parameters in individuals undergoing total hip arthroplasty. Forty-four individuals with hip osteoarthritis were included in current study. Individuals were randomized as study group (n=23) and control group (n=21) by drawing lots. Individuals in the study group were followed up with a personalized home-based exercise program for 6 weeks. Individuals in the control group were followed up with an exercise training brochure. The exercise program of the individuals in the study group was checked at two-week intervals and adjustments were made in the exercise program. All individuals were evaluated before the operation, 2 weeks after the operation, and 12 weeks after the operation, and their data were recorded. Range of motion was measured with an inclinometer, muscle strength was measured with a hand dynamometer, joint position sense was measured with a target angle test, pain was measured with a visual pain scale, leg length was measured with a tape measure, and finally, the Q angle was measured with a goniometer. In addition to these,Tampa kinesiophobia scale, Oxford hip score and international physical activity scale were used. Timed up-and-go test was used to evaluate functional performance. Foursquare step test was used to evaluate balance, and finally, tetrax posturography device was used to evaluate postural control.

DETAILED DESCRIPTION:
The aim of this study was to examine the patients who underwent Total Hip Arthroplasty surgery with the diagnosis of hip osteoarthritis.

Home-based exercise program given individually under the control of a physiotherapist is effective in reducing pain.

related factors (joint range of motion, muscle strength, kinesiophobia, physical activity), To investigate its effect on functional status, balance and postural control.

ELIGIBILITY:
Inclusion Criteria:

* Having surgery with a diagnosis of osteoarthritis
* Cases have unilateral hip osteoarthritis
* Not having received physical therapy in the 6 months before the surgery
* Total hip arthroplasty surgery should only be performed on posterior or posterolateral done with initiative

Exclusion Criteria:

* Presence of Dementia, Neurological Deficit
* Having other diseases that may affect balance (vertigo, previous CVO, neuropathy, epilepsy)
* Being on medication that may affect balance (antidepressants, antiepileptics, antipsychotics)
* Individuals who use alcohol heavily
* End stage organ failure
* Cancer patients under active treatment (except those in remission

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
OXFORD HİP SCORE | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  The Oxford Hip Score consists of 12 questions asking patients to describe their hip pain and function during the past 4 weeks. Each item uses a 5-point response scale with values from 0 to 4. An overall score is created by summing the responses to each of the 12 questions. The total score can range from 0 to 48 (most recent scoring system), where 0 is the worst possible score, indicating severe hip problems, and 48 is the best score, suggesting excellent hip function
TAMPA SCALE FOR KINESİOPHOBİA | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  It is a scale consisting of 17 questions created to measure fear of injury. The scale includes injury/re-injury and fear-avoidance parameters in work-related activities.A 4-point Likert scoring on the scale (I strongly disagree
  1, I disagree 2, I agree 3, I completely agree 4) is used. Individuals receive a total score between 17-68. A high score on the scale indicates that the person has a high level of kinesiophobia. Scores over 37 points are interpreted as high kinesiophobia.
İNTERNATİONAL PHYSİCAL ACTİVİTY QUESTİONAİRE (SHORT FORM) | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  The short form records the activity of four intensity levels: 1) vigorous-intensity activity such as aerobics, 2) moderate-intensity activity such as leisure cycling, 3) walking, and 4) sitting. The original authors recommended the "last 7 day recall" version of the questionaire for physical activity surveillance.
JOİNT POSİTİON SENSE ERROR TEST | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  The range of motion in the hip flexion direction is determined to be tested as active movement and passive movement in the 30 ˚, 60 ˚ and 90 ˚ positions. Movement deviations from specified angles are recorded along with the degree of deviation. The joint position sense error increases with the amount of deviation from the anticipated angle.
FOUR SQUARE STEP TEST | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  It is a measurement of dynamic standing balance.Performance time is calculated for each individual. Prolonged performances indicate an absence of equilibrium.
THE TİMED UP and GO TEST | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  The timed up and go test measures in seconds the time it takes a subject to rise from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down. This test has been used to examine balance, gait speed, and functional ability that would be required for the performance of basic activities of daily living in older people.
Assessment of Hip Muscle Strength | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  A microFET®2 (Digital Hand-held Dynamometer, Hoggan Scientific, LLC; Salt Lake City, Utah) Hand-Held Dynamometer is going to used to measure muscle strength. Using the break test method, which reveals isometric muscle contraction during the muscle test, force is applied in the opposite direction until a joint movement occurred exceeding the maximum power applied with the dynamometer. The strength of the healthy and osteoarthritic hip muscles are evaluated with the patient in supine position. The measurements are recorded as Newton (N) units.
Assessment of Hip Joint Range of Motion | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  Individuals' hip joint range of motion will be evaluated using the Baseline Bubble® Inclinometer. Hip flexion and abduction active range of motion will be evaluated in the standing position, and hip rotations will be evaluated in the supine position. Decreased hip joint range of motion is a clinical precursor of hip osteoarthritis, characterized by pain and loss of function.
Assessment of Postural Control | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  To evaluate postural control, measurements will be made with a software-based static posturography device (Tetrax®, Sunlight Medical Ltd). Tetrax® consists of four independent platforms that measure vertical pressure changes from both toes and both heels, and a computer software that combines the digital data from this platform. The system can digitally record data from four different measurement platforms in a certain period of time and document it as visual and numerical values. While measuring, individuals place their bare feet on the platforms and stand comfortably in a quiet environment. Individuals hold their head and eyes open and closed. It is evaluated in 8 different positions using neck rotations. The software evaluates postural control by generating a stability index with a numerical value from all measurements.

SECONDARY OUTCOMES:
MEASURİNG LEG LENGTH DİSCREPANCY | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  Leg length will be recorded in cm by measuring the distance between the major trochanter and the medial malleolus with a 6 mm tape measure.
Q ANGLE | Prior to surgery, two weeks following surgery, and twelve weeks following surgery, the same measurements will be taken.
  The patients are placed in the supine position, and the axis between the tibial tubercle and the midpoint of the patella is measured along with the axis between the spina iliaca anterior superior and the midpoint of the patella. The angle value between these two axes is then recorded numerically. Goniometers are used to take measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis AM, Perruccio AV, Ibrahim S, Hogg-Johnson S, Wong R, Streiner DL, Beaton DE, Cote P, Gignac MA, Flannery J, Schemitsch E, Mahomed NN, Badley EM. The trajectory of recovery and the inter-relationships of symptoms, activity and participation in the first year following total hip and knee replacement. Osteoarthritis Cartilage. 2011 Dec;19(12):1413-21. doi: 10.1016/j.joca.2011.08.007. Epub 2011 Aug 18. PMID 21889596
- [Background] Pop T, Szymczyk D, Majewska J, Bejer A, Baran J, Bielecki A, Rusek W. The Assessment of Static Balance in Patients after Total Hip Replacement in the Period of 2-3 Years after Surgery. Biomed Res Int. 2018 Jan 4;2018:3707254. doi: 10.1155/2018/3707254. eCollection 2018. PMID 29511678
- [Background] Ometti M, Brambilla L, Gatti R, Tettamanti A, La Cava T, Pironti P, Fraschini G, Salini V. Capsulectomy vs capsulotomy in total hip arthroplasty. Clinical outcomes and proprioception evaluation: Study protocol for a randomized, controlled, double blinded trial. J Orthop. 2019 Sep 12;16(6):526-533. doi: 10.1016/j.jor.2019.09.020. eCollection 2019 Nov-Dec. PMID 31680746
- [Result] Trudelle-Jackson E, Emerson R, Smith S. Outcomes of total hip arthroplasty: a study of patients one year postsurgery. J Orthop Sports Phys Ther. 2002 Jun;32(6):260-7. doi: 10.2519/jospt.2002.32.6.260. PMID 12061707